CLINICAL TRIAL: NCT03481088
Title: "Comparative Evaluation of the Temporomandibular Joint Disc-condyle-fossa Relationship Following Functional Appliance Therapy in Skeletal Class II Division 2 Malocclusion in Adolescent Females : A Magnetic Resonance Imaging Study"
Brief Title: "Changes in TMJ by Twin Block Therapy in Skeletal Class II Div 2 Malocclusion in Adolescent Females : MRI Study"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kavita
Record Dates: First submitted 2018-03-03; First posted 2018-03-29 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2018-03

CONDITIONS: Class II Division 2 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Myofunctional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional appliance therapy (Other): All records, including MRI scans will be collected at three stages and will be traced for various angular and linear measurements to document the alterations within the condyle glenoid fossa complex.
  1. Stage- I (pre-treatment),
  2. Stage- II (after pre-functional therapy)
  3. Stage-III (After 6-8 months of functional appliance therapy that is after correction to Class I molar relation)
  Interventions: Procedure: Functional appliance therapy

INTERVENTIONS:
Procedure: Functional appliance therapy — All records, including MRI scans will be collected at three stages and will be traced for various angular and linear measurements to document the alterations within the condyle glenoid fossa complex.
  1. Stage- I (pre-treatment),
  2. Stage- II (after pre-functional therapy)
  3. Stage-III (After 6-8 months of functional appliance therapy that is after correction to Class I molar relation)
  Other Names: myofunctional therapy

SUMMARY:
It is a prospective descriptive study to evaluate TMJ disc-condyle-fossa relationship using MRI scan following functional appliance therapy in skeletal Class II Division 2 malocclusion in adolescent females.

All records, including MRI scans will be collected at three stages and will be traced for various angular and linear measurements to document the alterations within the condyle glenoid fossa complex

1. Stage- I (pre-treatment),
2. Stage- II (after pre-functional therapy)
3. Stage-III (After 6-8 months of functional appliance therapy that is after correction to Class I molar relation

DETAILED DESCRIPTION:
Angle's class II division 2 malocclusion is relatively rare. Its frequency lies between 1.5 and 5% of all occlusion in white western population while in north Indian population it is 5.8% Generally in Class II division 2 malocclusion mandibular denture is more distally placed in relation to maxillary denture, a compensating effect in this type of mandibular retrusion , which offsets some of the disharmony of the facial profile is that the chin point is usually very pronounced3. It has been stated that patients with skeletal class II division 2 malocclusion ,when compared with normal class I or class II division I subject have larger masticatory muscles that in addition are oriented in a more anterior direction. These characteristics results in significant differences regarding their mechanical advantage and magnitude of occlusal forces.5 Several investigators have also stated that the mandible is locked posteriorly in Angle's Class II division 2 malocclusion with deep bite and the treatment which unlocks the bite during an active growth period can allow the mandible to grow or be repositioned forward much more than if treatment of unlocking of a bite were not undertaken. In class II division 2 malocclusion the condyle is positioned posteriorly while the disk is positioned anteriorly in relation to glenoid fossa. The articular disc in Angle's class II Division 2 patients could take a relative protrusive position in comparison with the other Angle's classes of malocclusion .

Successful treatment of many orthodontic problems depends to a great extent on the amount of mandibular growth patients experience during treatment. Functional appliances have been used for nearly 100 years in an attempt to induce mandibular growth by changing muscle function and condyle glenoid fossa relationships. Several studies have shown that the treatment of skeletal Class II patients with functional appliances is more successful when initiated during the adolescent growth spurt.

MRI a multiplanar imaging technique, has the advantage of giving an accurate assessment of both the bony and the soft tissues.It has high sensitivity for visualization of position and configuration of disc . This technique is believed to be non-invasive, radiation free and gives more superior contrast resolution than any other imaging modality. Recent studies have shown that we can have greater confidence in MRI as diagnostic tool because of improved quality.

MATERIALS AND METHODS- It is a prospective descriptive study to evaluate TMJ disc-condyle-fossa relationship using MRI scan following functional appliance therapy in skeletal Class II Division 2 malocclusion in adolescent females.

The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopedics, PGIDS, in association with the Department of Radiology, PGIMS, and Department of Oral Radiology, PGIDS, Pt B. D. Sharma University of Health Sciences, Rohtak.

. Ethical clearance approved by institutional Ethics Committee,Post Graduate Institute of Dental Sciences

Source of data:- The sample size consists of 15 subjects who were selected from the patients attending regular OPD at the Department of Orthodontics and Dentofacial Orthopedics for orthodontic treatment.

TARGET SAMPLE SIZE Sample size on= 13 for present study Calculation based on effect size of 1.23 with standard deviation of 10.5 at 95% confidence interval and 80% power n=2.{Z( 1-α/2)+Z(1-β)} 2/ ∆2 To compansate for 10 % dropout the final sample size will be 15

. INFORMED CONSENT OF THE PATIENT AND AGREEMENT TO BE RANDOMISED A valid, informed written consent of the patient or parent/ guardian and an agreement to be randomized was obtained from the patient before registering the patient in this clinical study. Patient or parent/ guardian was informed about all the theoretical risks and benefits of the intervention under test.

INTERVENTION AND DESIGN OF STUDY The study sample will consist of 15 growing females with skeletal class II and Angle's Class II division 2 malocclusion indicated for functional appliance therapy using Twin Block appliance.

The patients attending the regular OPD at the Department of Orthodontics and Dentofacial Orthopedics will be screened to match the inclusion criteria. Lateral Cephalograms will be taken to assess CVMI stage and growth pattern. Skeletal Class II Div 2 adolescent females with growth phase CVMI stage 2-4 having average to horizontal growth pattern as assessed by SN-MP (Go-Gn) angle will be included in the study.

Following detailed clinical examination, cephalometric analysis and treatment planning , the patients who will be ready to receive treatment will undergo pre-treatment MRI of condyle-glenoid fossa complex,then these patients will be treated with pre-functional therapy to correct retroclined incisors. After this, MRI of the TMJ of all these patients will be taken, that is after unlocking of mandible. Then these patients will undergo functional appliance therapy to achieve class 1 occlusion for an average of 6-8 months. After that, post fuctional MRI of the TMJ of all the patients will be taken.

The MRI protocol will include T1 weighted (T1W) spin echo sequences (TR 450/TE 15/Fov 160*160 mm), Proton density weighted spin echo sequences (TR 1500/TE 30/Fov 150*150) in coronal oblique and sagittal oblique planes of 3 mm slice thickness with no interslice gap. All records, including MRI scans will be collected at three stages and will be traced for various angular and linear measurements to document the alterations within the condyle glenoid fossa complex.

1. Stage- I (pre-treatment),
2. Stage- II (after pre-functional therapy)
3. Stage-III (After 6-8 months of functional appliance therapy that is after correction to Class I molar relation ANGULAR AND LINEAR MEASUREMENTS The eminence angle and the sagittal disc position measured in relation to two reference lines: the posterior condylar line (PC line) and the Frankfurt Horizontal plane (FH Plane). The PC line to be drawn directly on the MRI scan, while the FH plane transferred from the lateral cephalogram to the MRI scan, according to the method given by Nebbe et al.

Transfer of FH plane Determination of long axis of the condyle will be done by two step circle center method by Nebbe et al.

ANGULAR MEASUREMENTS 1-2) The eminence angle and the coronal disc position will be evaluated by the method described by Chintakanon et al.

3) The sagittal disc position will be evaluated using PC line and FH plane as described by Chintakanon et al.

4) Sagittal condylar concentricity will be evaluated using the method described by Pullinger et al.

5) The glenoid fossa angle will be measured on the sagittal films as the angle between the tangents to the anterior and posterior slopes of the glenoid fossa.

LINEAR MEASUREMENTS 6) Condyle and glenoid fossa displacements: The position of the glenoid fossa, and that of the condyle, will be evaluated with respect to the centre of the external auditory meatus (c-EAM). by marking one point at the centre of condyle (c-CH) and the linear distance of the c-CH from the c-EAM will be evaluated as the shortest distance from the constructed FH perpendicular.

7) Distance between c-PGS (crest of the post-glenoid spine ) & c-EAM : One point will be marked at the crest of the post-glenoid spine (c-PGS) and the linear distance of the c-PGS from the c-EAM will be evaluated as the shortest distance from the constructed FH perpendicular.

8) Superior joint space will be measured from the shortest distance between the most superior point of the condyle and the most superior point of the mandibular fossa.

Statistical analysis:-The data recorded will be processed by standard statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients in active growth period.
* Skeletal Class II base with mandibular retrognathia.
* Angle's Class II Division 2 malocclusion.
* Low anterior facial height.
* Patients having average to Horizontal growth pattern

Exclusion Criteria:

* Patients with any internal derangement or pathology of TMJ.
* History of previous orthodontic interventions or systemic diseases affecting bone metabolism.
* Growth abnormality.
* Patient with any endocrinal disorder
* Bleeding disorders.
* Patients with facial asymmetry

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
MRI comparisons for TMJ condyle-disc and glenoid fossa changes like sagital concenticity in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  measured in percentage displacement of condyle in the glenoid fossa
MRI comparisons for eminence angle in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  measured in degrees, the angle of anterior slope of glenoid fossa in relation to Frankfurt Horizontal plane and Posterior Condylar line
MRI comparisons for sagittal disc position in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  measured in degrees from references from Frankfurt Horizontal plane and Posterior Condylar line.
MRI comparisons for Linear glenoid fossa displacement in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  measured in millimetres, distance from external auditary meatus to centre of condylar head and Posterior glenoid spine
MRI comparisons for glenoid fossa angle measured in degree in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  measured in degrees, angle between anterior slope and posterior slope of glenoid fossa
MRI comparisons for coronal disc position in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  .relative position on the equal tenths on condyle. Negative value represents the lateral side; Positive value represents the medial side.
MRI comparisons for Superior joint space in pretreatment prefunctional and postfunctional MRI. | 16-18 months
  measured in millimetres, distance between most superior point on glenoid fossa and superiormost point on condyle.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Negi, MDS student, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided
Aim of the study is to document the alterations within the condyle-glenoid fossa complex and the positional changes of the glenoid fossa in the cranium after active functional phase like sagittal concentricity, eminence angle, sagittal disc position,glenoid fossa angle and linear metric measurements
  To evaluate TMJ changes using MRI scan after pre-functional therapy, that is after unlocking of mandible.
  To compare the mandibular condyle disc-fossa relationship on Magnetic resonance imaging in adolescent female having Angle's Class II Division 2 malocclusion before and after twin block functional appliance therapy.